CLINICAL TRIAL: NCT07021196
Title: The ICT Based Prescription of Physical Activity for Oncology Patients at Their Home: the EASYDOM Trial
Brief Title: The ICT Based Prescription of Physical Activity for Oncology Patients at Their Home
Acronym: EASYDOM
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Alessandra Cuomo, Assistant Professor, Federico II University
Other Study IDs: FedericoIIU 224/2024
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- Patients affected by breast or prostatic cancer: Patients affected by breast or prostatic cancer eligible for adiuvant treatment

SUMMARY:
Study evaluating the efficacy of ICT-based prescription of physical activity in oncology patients

ELIGIBILITY:
Inclusion Criteria:

* Female patients affected by breast cancer eligible for adiuvant treatment
* Male patients affected by prostatic cancer eligible for adiuvant treatment

Exclusion Criteria:

* Active life stily before enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by breast or prostatic cancer eligible for adiuvant treatment
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
tollerance to exercise | 6 months
  10% increase in time of exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Naples, Italy